CLINICAL TRIAL: NCT03536819
Title: Radio-frequency Rejuvenation for Pelvic Floor and Vagina
Brief Title: RF Rejuvenation for Pelvic Floor and Vagina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO607404A
Record Dates: First submitted 2018-05-08; First posted 2018-05-25 (Actual); Results first posted 2020-10-29 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Symptoms Associated With Pelvic Floor Weakness

STUDY DESIGN:
Intervention Model Description: Subjects will receive the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Participants receive Votiva treatment
  Interventions: Device: Votiva

INTERVENTIONS:
Device: Votiva — The applicator uses radio-frequency energy to treat the vaginal canal

SUMMARY:
Evaluation of efficacy and safety of the Votiva RF system with the Forma V handpiece for vaginal treatments.

DETAILED DESCRIPTION:
This study will evaluate the effects of radiofrequency on pelvic floor strength and the change in associated symptoms through direct measurement and patient reporting. The patients will undergo two separate evaluation appointments then receive two treatments. One group will receive a sham treatment and the other will receive the treatment. The sham group will be offered treatment at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult females between the ages of 35-75, seeking treatments for pelvic floor relaxation syndrome or atrophic vaginitis, which include but are not limited to: pelvic floor laxity, decreased muscle contraction in the pelvic floor, urinary incontinence, sexual dysfunction.
* Participants must have an evaluation by the Pelvic Floor Physical Therapists. All participants must have a minimum of 30% below average reading on initial assessment of internal or external pelvic floor contraction in order to be included in the study.
* Negative PAP smear and pelvic exam done within last 1 year.
* The patients should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, (including the permission to use photography).
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other treatment methods in the treatment areas such surgeries,CO2 treatment, other radiofrequency treatments and fillers injections for the last 12 months and during the entire study period.

Exclusion Criteria:

* Internal defibrillator, pacemaker, bladder stimulator or any other implanted electrical device anywhere in the body
* Permanent metal implant in the treatment area
* History of pelvic floor radiation
* Any surgery in the treatment area in the last 3 months
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* Pregnancy and nursing
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes, thyroid dysfunction, polycystic ovary and hormonal virilization
* Any active condition in the treatment area, such as but not limited to open sores, psoriasis, eczema,vitiligo,herpes and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Diseases that may be stimulated by light, such as epilepsy, lupus and urticaria.
* Any other previous treatments in the vaginal or perineal area, such as CO2 laser or RF performed on the same area.
* Any surgical procedure in the vaginal area within the past 12 months.
* Recent tan from sun, sunbeds or chemicals or planned excessive sun exposure.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Kouris, MD, Principal Investigator — Midwest Plastic Surgery, 5201 S. Willow Springs Road, Suite 440 LaGrange, IL, 60525
Locations (1):
- Midwest Plastic Surgery, LaGrange, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] — Population: Only subjects that finished all visits were analyzed
  years
    number analyzed (Participants) | 15
    (all) | 51.8 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only subjects that finished all visits were analyzed
  Participants
    number analyzed (Participants) | 15
    Female | 15
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 18
  Black or African American | 1
  Hispanic or Latino | 1
Intentional muscle contraction using Biofeedback EMS [Mean (Standard Deviation); unit: mV] — EMS Biofeedback using a vaginal sensor for evaluation of Pelvic floor muscle strength. There is no signal normalization, this measurement tool is used to measure change in Pelvic Floor Muscle function.
  Pelvic floor muscle Contractions amplitude are measured in mV (microvolt)
  1. Peak internal Pelvic Floor Contractions (steadily higher scores demonstrate improvement) Population: Only subjects that finished all visits were analyzed
  mV
    number analyzed (Participants) | 15
    (all) | 9.69 (5.65)
Urinary Incontinence symptoms International Consultation on Incontinence Questionnaire ICIQ [Mean (Standard Deviation); unit: score on a scale] — ICIQ-Subjective assessment of efficacy on Urinary Incontinence symptoms using the International Consultation on Incontinence Questionnaire ( lower scores demonstrate improvement). The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. Scoring scale: 0-21. Population: Only subjects that finished all visits were analyzed
  score on a scale
    number analyzed (Participants) | 15
    (all) | 5.71 (3.53)
Female Sexual Function Index (FSFI) [Mean (Standard Deviation); unit: score on a scale] — FSFI - Subjective assessment of efficacy on sexual dysfunction symptoms, using the Female Sexual Function Index 2-36, increasing scores demonstrate improvement) Population: Only subjects that finished all visits were analyzed
  score on a scale
    number analyzed (Participants) | 15
    (all) | 23.10 (6.50)
Pelvic Floor Impact Questionnaire (PFIQ-7) [Mean (Standard Deviation); unit: score on a scale] — PFIQ-7 - Subjective assessment of quality of life change using Pelvic Floor Impact Questionnaire, 0-300, lower scores demonstrate improvement Population: Only subjects that finished all visits were analyzed
  score on a scale
    number analyzed (Participants) | 15
    (all) | 18.73 (25.67)
Questionnaire for Urinary Incontinence Diagnosis (QUID) [Mean (Standard Deviation); unit: score on a scale] — QUID - Questionnaire for Urinary Incontinence Diagnosis. QUID- scaled 0-15, larger values indicating worse UI. Population: Only subjects that finished all visits were analyzed
  score on a scale
    number analyzed (Participants) | 15
    (all) | 9.67 (6.74)
PISQ-12 Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire [Mean (Standard Deviation); unit: score on a scale] — PISQ-12 short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire . PISQ12 score calculator evaluates sexual function in women with urinary incontinence or pelvic organ prolapse. Score 0-48. Higher number demonstrate improvement. Population: Only subjects that finished all visits were analyzed
  score on a scale
    number analyzed (Participants) | 15
    (all) | 32.67 (5.19)
Pelvic Floor Distress Inventory (PFDI-20) [Mean (Standard Deviation); unit: score on a scale] — PFDI-20. Pelvic Floor Distress Inventory . The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is the short-form version of the Pelvic Floor Distress Inventory (PFDI). It is a health-related quality of life questionnaire for women with pelvic floor conditions. The PFDI-20 is comprised of 3 scales, which include the Urinary Distress Inventory-6 (UDI-6), Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8. Score 0-300 Lower score demonstrate improvement. Population: Only subjects that finished all visits were analyzed
  score on a scale
    number analyzed (Participants) | 15
    (all) | 84.93 (55.08)

OUTCOME MEASURES:

1. Primary Outcome: Effect of RF on Pelvic Floor Measured by Intentional Muscle Contraction Using Biofeedback EMS
Description: There is no signal normalization, this measurement tool is used to measure change in Pelvic Floor Muscle function.
  Pelvic floor muscle Contractions amplitude are measured in mV (microvolt)
  1. Peak internal Pelvic Floor Contractions (steadily higher scores demonstrate improvement)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Treatment
Number analyzed (Participants) | 15
mV | 13.13 (5.96)

2. Primary Outcome: Recording of Adverse Events (Safety)
Description: Observation, assessment and recording of reactions
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 15
participants | 0

3. Secondary Outcome: Evaluate Urinary Symptoms Associated With Pelvic Floor Weakness
Description: ICIQ-Subjective assessment of efficacy on Urinary Incontinence symptoms using the International Consultation on Incontinence Questionnaire ( lower scores demonstrate improvement). The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. Scoring scale: 0-21.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale | 3.53 (3.36)

4. Secondary Outcome: Evaluate Sexual Dysfunction Symptoms Associated With Pelvic Floor Weakness
Description: FSFI - Subjective assessment of efficacy on sexual dysfunction symptoms, using the Female Sexual Function Index 2-36, increasing scores demonstrate improvement)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale | 26.19 (6.53)

5. Secondary Outcome: Evaluate Quality of Life Symptoms Associated With Pelvic Floor Weakness
Description: PFIQ-7 - Subjective assessment of quality of life change using Pelvic Floor Impact Questionnaire, 0-300, lower scores demonstrate improvement
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale | 12.7 (21.57)

6. Secondary Outcome: Evaluate Urinary Incontinence Symptoms
Description: QUID - Questionnaire for Urinary Incontinence Diagnosis. QUID- scaled 0-15, larger values indicating worse UI.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale | 6.87 (5.26)

7. Secondary Outcome: Evaluate Sexual Function Associated With Pelvic Floor Weakness
Description: PISQ-12 short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire . PISQ12 score calculator evaluates sexual function in women with urinary incontinence or pelvic organ prolapse. Score 0-48. Higher number demonstrate improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale | 35.6 (6.95)

8. Secondary Outcome: Evaluate Quality of Life With Pelvic Floor Conditions
Description: PFDI-20. Pelvic Floor Distress Inventory . The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is the short-form version of the Pelvic Floor Distress Inventory (PFDI). It is a health-related quality of life questionnaire for women with pelvic floor conditions. The PFDI-20 is comprised of 3 scales, which include the Urinary Distress Inventory-6 (UDI-6), Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6), and the Colorectal-Anal Distress Inventory-8. Score 0-300 Lower score demonstrate improvement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 15
score on a scale | 77.64 (43.84)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03536819/Prot_006.pdf
  • Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03536819/SAP_007.pdf
  • Informed Consent Form (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03536819/ICF_008.pdf